CLINICAL TRIAL: NCT00787293
Title: A Multi-center Study of the Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty System to Reduce Mitral Valve Regurgitation in Patients With Heart Failure
Brief Title: Study of Safety and Efficacy of the Percutaneous Reduction of Mitral Valve Regurgitation in Heart Failure Patients
Acronym: PTOLEMY-2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Company ended operations January 2011
Sponsor: Viacor (Industry)
Collaborators: Duke University (Other); Medifacts International Corporation (Industry)
Responsible Party: Katharine M Stohlman, Viacor, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-010P
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Heart Failure; Mitral Regurgitation
Keywords: Heart Failure; Mitral Regurgitation; Percutaneous; Coronary sinus
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patient is screened for study and given baseline assessments. Pending fulfillment of study eligibility criteria, patient is implanted with PTMA system.
  Interventions: Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant

INTERVENTIONS:
Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant — Percutaneous assessment from right or left subclavian vein, with PTMA implant in the coronary sinus, great cardiac vein, anterior interventricular vein.

SUMMARY:
Improvement in heart failure with moderate to severe mitral regurgitation using a percutaneously delivered implantable device.

ELIGIBILITY:
Inclusion Criteria:

* Functional MR 2+ - 4+
* Symptomatic heart failure, NYHA Class II to IV
* LVEF > 25% or < 50% OR dilated mitral annulus > 30mm

Exclusion Criteria:

* MR of organic origin
* Severe mitral leaflet tethering
* History of MI or PCI within 60 days of study procedure
* Inability to walk a minimum of 100 meters in 6 minutes
* Significant left main stenosis or proximal circumflex stent
* Indication of non-patent CSO or discontinuous CS-GCV-AIV
* Bi-ventricular with leads in CS or other devices impeding device placement
* Severe aortic valvular disease
* Chronic corticosteroid use other than < 20mg prednisone for arthritis
* Significant co-morbidities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Freedom from MACE at 30 days post-procedure and quantitative MR reduction at 6 months | 30 days to 6 months

SECONDARY OUTCOMES:
% of patients experiencing procedure or device-related adverse events | 30 days to 6 months
Technical procedural success: % of patients maintaining a reduction of mitral annulus A/P dimension, sustained MR reduction, and decrease in left ventricular dimensions to specified degrees | 6 months
Clinical status: % of treated patients exhibiting improvements in defined QoL parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sack, Md, PhD, Principal Investigator — Klinikum Schwabing, Staedtisches Klinikum Muenchen GmbH; Rainer Hoffmann, MD, Principal Investigator — R-WTH Universitätsklinikum Aachen
Locations (13):
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis Cardiovasculair Ondrezoek Aalst, Aalst
  - Centre Hospitalier Universitaire de Liège, Liège
- Institut Klinicke a Experimentalni Mediciny, Prague, Czechia
- Germany (7):
  - Rheinisch-Westfalische Technische Hochschule Universitaetsklinikum Aachen, Aachen
  - Herz-und Diabeteszentrum Nordrhein-Westfalen / Ruhr University of Bochum, Bad Oeynhausen
  - Universitaet Duisburg-Essen Westdeutsches Herzzentrum Universitaetsklinikum Essen, Essen
  - CardioVascular Center Frankfurt Sankt Katharinen, Frankfurt
  - Albert-Ludwigs-Universitat Freiburg Mediziniche Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Städtische Klinikum Karlsruhe GmbH, Karlsruhe
  - Klinikum Schwabing Städtisches Klinikum München GmbH, München
- Netherlands (2):
  - Thoraxcentrum Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Hôpital Universitaire de Genève, Geneva, Switzerland

REFERENCES:
- [Background] Fukuda S, Gillinov AM, Liddicoat JR, Saracino G, Hayase M, Cohn WE, Schneider CW, Shiota T. Maintenance of geometric alterations associated with percutaneous mitral valve repair: real-time three-dimensional echocardiographic assessment in an ovine model. J Heart Valve Dis. 2008 May;17(3):276-82. PMID 18592924
- [Background] Daimon M, Gillinov AM, Liddicoat JR, Saracino G, Fukuda S, Koyama Y, Hayase M, Cohn WE, Ellis SG, Thomas JD, Shiota T. Dynamic change in mitral annular area and motion during percutaneous mitral annuloplasty for ischemic mitral regurgitation: preliminary animal study with real-time 3-dimensional echocardiography. J Am Soc Echocardiogr. 2007 Apr;20(4):381-8. doi: 10.1016/j.echo.2006.08.029. PMID 17400117
- [Background] Dubreuil O, Basmadjian A, Ducharme A, Thibault B, Crepeau J, Lam JY, Bilodeau L. Percutaneous mitral valve annuloplasty for ischemic mitral regurgitation: first in man experience with a temporary implant. Catheter Cardiovasc Interv. 2007 Jun 1;69(7):1053-61. doi: 10.1002/ccd.21186. PMID 17525965
- [Background] Daimon M, Shiota T, Gillinov AM, Hayase M, Ruel M, Cohn WE, Blacker SJ, Liddicoat JR. Percutaneous mitral valve repair for chronic ischemic mitral regurgitation: a real-time three-dimensional echocardiographic study in an ovine model. Circulation. 2005 May 3;111(17):2183-9. doi: 10.1161/01.CIR.0000163547.03188.AC. Epub 2005 Apr 25. PMID 15851597
- [Background] Liddicoat JR, Mac Neill BD, Gillinov AM, Cohn WE, Chin CH, Prado AD, Pandian NG, Oesterle SN. Percutaneous mitral valve repair: a feasibility study in an ovine model of acute ischemic mitral regurgitation. Catheter Cardiovasc Interv. 2003 Nov;60(3):410-6. doi: 10.1002/ccd.10662. PMID 14571496